CLINICAL TRIAL: NCT03607903
Title: A Randomized, Double Blind, Placebo-controlled, Double-dummy Study to Assess Microneedle Delivery in Comparison to Subcutaneous Injection of Adalimumab in Healthy Volunteers
Brief Title: Adalimumab Microneedles in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Leiden University Medical Center (Other); Leiden Academic Center for Drug Research, the Netherlands (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CHDR1807
Record Dates: First submitted 2018-06-08; First posted 2018-07-31 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Pain; Injection Site
Keywords: intradermal; adalimumab; microneedle; subcutaneous; healthy volunteers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a double blind, placebo controlled, double-dummy study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double blind. Investigator, study staff, and subjects, are blinded until study closure. Investigational drug and matching placebo are indistinguishable and will be packaged similarly. Injection site assessments will be performed by (a) study-independent physician(s). The study physician will administer the injection, thus unblinded to type of injection. This physician will not reveal the route of administration to others. The investigator receives sealed emergency codes to be broken in case of emergency situations. If the identity of study drug administered needs to be known to manage the subject's condition i.e., in case of a medical emergency or in the case a SUSAR occurs, the treatment emergency code for that subject may be broken and the study drug identified. All such occurrences should be documented in the study file. Just prior to database lock unused emergency code labels will be checked and a statement that all are intact (or not) is made on database lock form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Subcutaneous adalimumab and placebo (Active Comparator): adalimumab SC (40 mg in 0.4 mL) and saline ID (0.9%, 0.4 mL)
  Interventions: Biological: Adalimumab SC; Other: Saline ID
- PLacebo and subcutaneous adalimumab (Active Comparator): saline ID (0.9%, 0.4 mL) and adalimumab SC (40 mg in 0.4 mL)
  Interventions: Biological: Adalimumab SC; Other: Saline ID
- Placebo and intradermal adalimumab (Experimental): saline SC (0.9%, 0.4 mL) and adalimumab ID (40 mg in 0.4 mL)
  Interventions: Biological: Adalimumab ID; Other: Saline SC
- Intradermal adalimumab and placebo (Experimental): adalimumab ID (40 mg in 0.4 mL) and saline SC (0.9%, 0.4 mL)
  Interventions: Biological: Adalimumab ID; Other: Saline SC

INTERVENTIONS:
Biological: Adalimumab ID — Adalimumab intradermal using MicronJet600 microneedle from NanoPass
  Arms: Intradermal adalimumab and placebo; Placebo and intradermal adalimumab
Biological: Adalimumab SC — Adalimumab subcutaneous using regular needle
  Arms: PLacebo and subcutaneous adalimumab; Subcutaneous adalimumab and placebo
Other: Saline ID — Saline intradermal using MicronJet600 microneedle from NanoPass
  Arms: PLacebo and subcutaneous adalimumab; Subcutaneous adalimumab and placebo
Other: Saline SC — Saline subcutaneous using regular needle
  Arms: Intradermal adalimumab and placebo; Placebo and intradermal adalimumab

SUMMARY:
Adalimumab (Humira, AbbVie) is a highly effective treatment for a variety of auto-immune/auto-inflammatory diseases including juvenile idiopathic arthritis (JIA). Adalimumab works by binding to tumor necrosis factor alpha (TNF), hereby preventing its interaction with the TNF receptor. In the presence of complement, adalimumab can also lyse TNF-expressing cells.

Adalimumab is administered via subcutaneous injection, which has the major drawback of being perceived as unpleasant and painful, especially during long term use for both adults and children. As subcutaneous administration may therefore eventually jeopardize treatment adherence, there is a clear need for less invasive alternatives to administer highly effective biological drugs such as adalimumab.

Microneedles may be a potential alternative for invasive drug administration. Microneedles are currently widely investigated for the administration of various vaccines. The experience with administration of biological drugs is rather limited. The sparse available data suggests similar pharmacokinetics of adalimumab when administered either subcutaneous or intradermal in healthy volunteers. Moreover, the first studies report good tolerability of microneedles. However, no systematic studies have been performed yet i) to investigate pain, acceptability, and local tolerability for intradermal versus subcutaneous adalimumab administration ii) to evaluate safety, PK and immunogenicity for intradermal versus subcutaneous adalimumab and iii) to explore the usability of optical coherence tomography, clinical photography, thermal imaging and laser speckle contrast imaging in the evaluation of intradermal injections.

This study will directly compare the pain perception and hence acceptability of a single dose (40 mg) of adalimumab administered subcutaneously (SC) versus intradermally (ID) via microneedles in healthy adult volunteers. Furthermore, the pharmacokinetic profile, pharmacodynamics, the immunogenicity and the tolerability will be assessed. This study will enable bridging to a future study in children and adolescents with JIA, in which the suitability of microneedles for the administration of adalimumab in pediatric patients will be examined. The overarching aim of these studies is to make administration of biologicals in children as pain free as possible.

DETAILED DESCRIPTION:
Objective(s)

1. To evaluate the pain, acceptability and local tolerability of intradermal microneedle injection compared to subcutaneous injection in healthy volunteers.
2. To evaluate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of adalimumab after administration using microneedles versus subcutaneous injection in healthy volunteers.
3. To explore the usability of optical coherence tomography, clinical photography, laser speckle contrast imaging, and thermal imaging in the evaluation of intradermal injections.

Definitions Method: ID or SC injection Compound: adalimumab or saline Treatment: combination of method and compound Arm: sequence of treatments

Design This is a double blind, placebo controlled, double-dummy study. The study physician will administer the injection and is thus unblinded to the type of injection. All injection site assessments will be performed by (a) study independent member of the clinical staff.

Sterile saline injection will be used as a negative control. Subjects will receive an injection with both sterile saline (SC or ID) and adalimumab (SC or ID). Subjects will be randomized to one of the four arms:

1A) adalimumab SC and saline ID

1. B) saline ID and adalimumab SC
2. A) saline SC and adalimumab ID

2B) adalimumab ID and saline SC

The maximum duration between treatments will be 5 minutes.

After a single dose of adalimumab, pharmacokinetic, pharmacodynamics, tolerability and immunogenicity data will be collected and monitored for a total of 70 days post dose, as the half-life of adalimumab after subcutaneous injection in adults is approximately two weeks.

Investigational drug/device combination In children, adalimumab is commonly used in a dose of 40 mg SC every two weeks (1). For adults with rheumatoid arthritis the same dose is used (2). It was therefore chosen to administer adalimumab in a single dose of 40 mg in 0.4 mL either subcutaneously or intradermally in the upper thigh. For saline injection the same volume will be used.

For intradermal administration, the MicronJet600 (NanoPass Technologies) will be used (hereafter referred to as microneedle). This CE-marked microneedle consists of an array of three hollow pyramid-shaped microneedles with a length of 600 micrometer (3).

Subjects / Groups A total of 24 healthy subjects (N=6 per arm and N=12 per treatment (Adalimumab SC, Adalimumab ID, Saline SC, Saline ID).

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following inclusion criteria at screening:

1. Healthy male / female subjects, 18 to 45 years of age, inclusive at screening;
2. Good health, based upon the results of medical history, physical examination, vital signs, ECG, and laboratory profiles of both blood and urine;
3. Body mass index (BMI) between 18 and 30 kg/m2, inclusive at screening, and with a minimum weight of 50 kg;
4. Willing to practice an approved method of birth control and not breastfeeding throughout the study and for five months after study drug administration, as advised in the drug formulary (2). If the trial subject is female, surgical sterilization or postmenopausal status for >1 year will satisfy this requirement. All female subjects are required to have a negative pregnancy test at screening and at baseline (pre-dose);
5. Fitzpatrick skin type I-II (Caucasian type);
6. Suitable site for intradermal injection on the legs, as assessed by the investigator;
7. Able and willing to provide written informed consent.

Exclusion Criteria:

Eligible subjects must meet none of the following exclusion criteria at screening:

1. Immune-compromised (known or expected immune deficiency, disease, or use of medication that may affect the immune system);
2. Diagnosed with tuberculosis (TB, as per positive skin test [Mantoux] or interferon gamma release assay), or history of TB, or latent TB, or recent contact with TB (patient); having travelled to countries where TB is endemic within eight weeks of planned drug administration or planning to travel to countries where TB is endemic from the moment of drug administration until three months after the end of the study;
3. Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug (including adalimumab);
4. History of chronic infection, or infections within the past two years requiring hospitalization or administration of intravenous antibiotics;
5. Receipt of any live vaccination within three months prior to study drug administration, or intention to undergo live vaccinations from the moment of drug administration until four months after the end of study;
6. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening;
7. Evidence of any active or chronic disease (hematologic, renal, hepatic, cardiovascular, neurologic, endocrinal, gastrointestinal, oncologic, pulmonary, immunologic, or psychiatric disorder) or condition that could interfere with, or for which the treatment of might interfere with the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator (following a detailed medical history, physical examination, vital signs (systolic and diastolic blood pressure, and body temperature) and ECG). Minor deviations from the normal range may be accepted, if judged by the investigator to have no clinical relevance;
8. History of abuse of addictive substances (alcohol, illegal substances) or current use of more than 21 units alcohol per week, drug abuse, or regular user of sedatives, hypnotics, tranquillisers, or any other addictive agent;
9. Consumption of alcohol within the 48-hour period prior to study drug administration;
10. Smoke more than 10 cigarettes per day prior to screening or use tobacco products equivalent to more than 10 cigarettes per day and/or unable to abstain from smoking whilst in the unit;
11. Positive screen for recreational drugs or alcohol;
12. Is demonstrating excess in xanthine consumption (more than eight cups of coffee or equivalent per day);
13. Unlikely to comply with the study protocol and/or to complete the study or required study procedures, including being unlikely or unable to return for follow-up visits;
14. Use of any medication (prescription or over-the-counter (OTC) within 14 days of study drug administration, or use of herbal supplements, dietary supplements or multivitamins within 7 days of study drug administration or less than five half-lives (whichever is longer), or receipt of any drug by injection within 30 days of study drug administration, with the exception of contraceptives, hormonal replacement therapies, and paracetamol (up to 4g/day). Other exceptions will only be made if the rationale is clearly documented by the investigator;
15. Donation of over 500 mL of blood within three months prior to screening or donation of plasma within 14 days prior to screening;
16. Previous exposure to any biological;
17. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times in the past year;
18. Excessive sun exposure of the injection site area within 3 weeks of enrollment;
19. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive adalimumab or otherwise participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Amount of pain | 7 weeks
  Pain will be measured using a standard 100 points visual analogue scale (0: no pain, 100: extreme pain).
  Insertion, injection and post-injection pain will be assessed separately.
Adalimumab pharmacokinetics | 10 weeks
  Individual serum adalimumab concentrations will be plotted versus time per individual.
Anti-adalimumab antibodies | 10 weeks
  All subjects who received study medication will be monitored for serum anti-adalimumab antibodies.
Ex vivo cytokine levels | 10 weeks
  Ex vivo whole blood challenge will be performed to assess the effect of adalimumab on the release of cytokines by circulating immune cells and activation of these cells. Whole blood will be stimulated with 2ng/mL lipopolysaccharide and 25 ug/mL aluminium ydroxide for 24 hours at 37 degrees Celsius, 5% carbon dioxide. Culture supernatants will be assayed for release of pro-inflammatory cytokines including tumor necrosis factor alpha, interleukin 6, interleukin 1 beta, interleukin 8, and interferon gamma.
Amount of pain | 7 weeks
  Pain will be measured using Dutch version of the faces pain scales revised (0-2-4-6-8-10, 0: no pain, 10: very much pain).
  Insertion, injection and post-injection pain will be assessed separately.

SECONDARY OUTCOMES:
Preference for subjects for either injection (SC versus ID) | 2 days
  Subjects will be asked multiple choice questions on the acceptability of both injections.
Number of injection site reactions | 10 weeks
  Injection site assessment for the following:
  Pain (grade 1/2/3) Tenderness (grade 1/2/3) Pruritus (grade 1/2/3) Erythema (absent/present) Induration (grade 1/2/3) Blister (absent/present) Ulceration (absent/present) Necrosis (absent/present) Ecchymosis (absent/present) If any of these signs or symptoms is present, it is regarded an injection site reaction.
Number of (serious) adverse events per treatment arm | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, RPh PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
CHDR will provide NanoPass with a written report summarizing the results of the Clinical Study such as the publication or manuscript, including but not limited to, promptly sharing any severe or potentially reportable safety or adverse event potentially related to the MicronJet600.